CLINICAL TRIAL: NCT04694547
Title: Ketogenic Diet Survey in GSDV
Brief Title: Ketogenic Diet Survey in Patients With McArdle Disease (GSDV)
Status: Completed | Type: Observational
Sponsor: Nicoline Løkken (Other)
Responsible Party: Sponsor-Investigator, Nicoline Løkken, Principal Investigator, MD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: Ketogenic diet survey in GSDV
Record Dates: First submitted 2020-10-05; First posted 2021-01-05 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: McArdle Disease
MeSH Terms: conditions — Glycogen Storage Disease Type V

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: There is no intervention, as this is a survey study — Survey

SUMMARY:
The purpose of this survey is to report experiences with variants of a ketogenic diet in a group of individuals diagnosed with McArdle disease (glycogen storage disease type V). Further more the survey will report on physical activity, fatigue, sleep and quality of life in this cohort.

DETAILED DESCRIPTION:
Currently, there is no satisfactory treatment for McArdle disease. The limitation in people with McArdle disease is due to a limited availability of energy in the muscle due to affected carbohydrate metabolism. A key element in improving muscle function is therefore to introduce alternative energy sources. Ketone bodies are a well-known source of energy for both brain and muscle. Ketone bodies are produced during fasting or when following a ketogenic diet. A ketogenic diet is a diet high in fat and low in carbohydrates. The classic ketogenic diet contains up to 90% fat, but there are several alternative diets with less fat, including a modified ketogenic diet, Atkins diet, LCHF (low carb high fat), OMAD (one meal a day) and more. This survey will collect information on all variations. The rationale for a ketogenic diet for persons with McArdle disease makes good sense in theory, as the diet would contribute with a new source of energy (ketone bodies) independent of the affected carbohydrate breakdown. However, evidence is sparse on whether the diet actually works. The primary purpose of this survey is to report experiences with variants of the ketogenic diet in a group of individuals diagnosed with McArdle disease. Secondarily this survey will collect information on physical activity, fatigue, sleep and quality of life in this cohort

ELIGIBILITY:
Inclusion Criteria:

* Verified GSDV diagnosis

Exclusion Criteria:

* Age under 18 years

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: McArdle disease
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Questions on experiences with a ketogenic diet | Baseline
  Survey
IPAQ (INTERNATIONAL PHYSICAL ACTIVITY QUESTIONNAIRE) short form | Baseline
  Survey
MFI-20 (MULTIDIMENSIONAL FATIGUE INVENTORY) | Baseline
  Survey
ISI (insomnia severity index) | Baseline
  Survey
MGQOL 15 score (Myasthenia Gravis Quality Of Life) | Baseline
  Survey

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen Neuromuscular Center, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Reason SL, Lokken N, Voermans N. International patient group harnesses social media to help inform rare disease research: use of a low carbohydrate ketogenic diet in McArdle disease. Curr Opin Endocrinol Diabetes Obes. 2021 Oct 1;28(5):441-445. doi: 10.1097/MED.0000000000000663. PMID 34269712